CLINICAL TRIAL: NCT05695118
Title: Analysis of the Prognostic Correlation Between Body Composition Analysis and Fatty Liver Progression in Patients With Fatty Liver Using Low-dose CT
Brief Title: Body Composition and Fatty Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUH-2022-3238
Record Dates: First submitted 2022-12-24; First posted 2023-01-23 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Fatty Liver
Keywords: CT
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- non-contrast low-dose abdomen CT (Experimental): non-contrast low-dose abdomen CT (target effective dose: < 1.5 mSv). CT based body composition analysis is performedd with commercially available automatic segmentation software (DeepCatch, Medical IP, South Korea).
  Interventions: Diagnostic Test: Non-contrast low-dose abdomen CT; Diagnostic Test: Fibroscan; Diagnostic Test: bioelectrical impedance analysis (BIA)

INTERVENTIONS:
Diagnostic Test: Non-contrast low-dose abdomen CT — target effective dose: < 1.5 mSv It is performed twice in 6-month interval.
Diagnostic Test: Fibroscan — Fibroscan is performed within a week of low-dose CT. It is used as a reference standard of hepatic fibrosis and steatosis.
Diagnostic Test: bioelectrical impedance analysis (BIA) — BIA test is performed on the same day of low-dose CT. Commercially available model (Inbody 270) is used.
  Other Names: Inbody test (commercial name)

SUMMARY:
This study investigates relationship between fatty liver prognosis and body composition analysis result based on non-contrast low dose CT in patients with fatty liver disease.

ELIGIBILITY:
Inclusion Criteria:

* metabolic dysfunction-associated fatty liver disease (fatty liver with overweight/obesity, or type II DM or other metabolic dysfunction)
* or non-alcoholic fatty liver disease with liver function test abnormality
* signed informed consent

Exclusion Criteria:

* chronic hepatitis B or C
* other disease related to fatty liver such as glycogen storage disease, lipodystrophy, familial combined hyperlipidemia, hypobetalipoproteinemia, Weber-Christian syndrome or abetalipoproteinemia
* on medication related to hepatic steatosis (tamoxifen, steroid, valproic acid, methotrexate, amiodarone)
* diabetes after pancreatectomy
* history of total parenteral nutrition in 6 months
* pregnancy or nursing mother

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
relationship between body composition analysis result from CT and liver fat fraction | 6 month after CT acquisition
  relationship between visceral fat volume fraction (obtained from CT analysis using automatic body segmentation, unitless (visceral fat fraction = visceral fat volume/total body volume)) and CAP value of fibroscan

SECONDARY OUTCOMES:
ratio of appropriate non-contrast low dose abdomen CT acquisition & analysis | 6 month after CT acquisition
  Number of CT scan with effective dose < 1.5 mSv AND successful automatic body composition analysis (without manual editing) divided by total number of CT scan
relationship between body composition analysis result from CT and hepatic fibrosis | 6 month after CT acquisition
  relationship between visceral fat volume fraction (CT analysis using automatic body segmentation, unitless (visceral fat fraction = visceral fat volume/total body volume)) and liver stiffness value of fibroscan
agreement between body composition analysis result from CT and bioelectrical impedance analysis (Inbody test) | 6 month after CT acquisition
  agreement of visceral fat, subcutaneous fat, muscle amount between CT based body composition and Inbody test results

OTHER OUTCOMES:
incidence of incidental finding | 6 month after CT acquisition
  incidentally detected findings on low-dose abdomen CT

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Professor
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No